CLINICAL TRIAL: NCT06303583
Title: Neoadjuvant Chemoradiotherapy Followed by Sequential Immunotherapy for Thoracic Esophageal Squamous Cell Carcinoma
Acronym: CRIS
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qiu Guoqin (Other)
Responsible Party: Sponsor-Investigator, Qiu Guoqin, Chief Physician, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB- 2022-213
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Neoadjuvant; chemoradiotherapy; tislelizumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Carboplatin; tislelizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IO (Experimental): chemoradiotherapy sequential tislelizumab
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: tislelizumab; Radiation: radiotherapy

INTERVENTIONS:
Drug: paclitaxel — paclitaxel, 50 mg/m2, QW*5
Drug: carboplatin — area under the curve of2mg/mL/min, QW*5
Drug: tislelizumab — 200mg Q3W, 2cycles
Radiation: radiotherapy — 41.4Gy in 23 fractions

SUMMARY:
The purpose of study is to investigate the safety and efficacy of sequential immunotherapy with neoadjuvant chemoradiotherapy for esophageal cancer

DETAILED DESCRIPTION:
This is a single-arm, phase Ib study. Eligibility criteria include histologically confirmed ESCC and clinical T3-4aN0M0 or T2-4aN+M0 (AJCC/UICC 8). Patients received neoadjuvant radiotherapy (41.4Gy in 23 fractions) with concurrent chemotherapy (paclitaxel, 50 mg/m2, carboplatin area under the curve of 2mg/mL/min, QW*5). Then followed by two cycles of tislelizumab (200mg, Q3W). The primary endpoint was the pathological complete response (pCR) rate and safety.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75.
* Histology confirmed thoracic esophageal squamous cell carcinoma.
* ECOG ps 0 to 1.
* Resectable or potentially resectable T2-4aN0 or T1-4aN+ patients (AJCC/UICC Clinical Staging of Esophageal squamous cell Carcinoma, 8th edition (cTMN)).
* Length of esophageal lesions <8cm.
* There were no surgical contraindications.
* Neutrophil count ≥1.5*109/L, platelet count ≥10.0*109/L, hemochrome ≥9g/dL; Serum creatinine ≤1.5 times the upper limit of normal value; Bilirubin ≤1.5 times the upper limit of normal value, AST, ALT, AKP≤2.5 times the upper limit of normal value.
* BMI acuity 18.5 kg/m2.
* Informed notification and signed informed consent.

Exclusion Criteria:

* Cervical esophageal cancer (upper part of the lesion in the cervical esophagus). Multifocal esophageal carcinoma, lesion length >8cm.
* Trachea and aorta were invaded (Annex 5).
* Hoarseness caused by the tumor.
* Esophageal fistula.
* Lymph node metastasis in the neck and periceliac artery (AJCC/UICC 8th edition esophageal/esophagogastric junction region lymph node division 1 and 20).
* A history of active autoimmune disorders or syndromes requiring treatment with systemic steroids or immunosuppressants (except for vitiligo or cured childhood asthma/allergies who do not require any intervention in adulthood; Autoimmune hypothyroidism treated with a stable dose of thyroid replacement hormone).
* She is on hormonal or immunosuppressive therapy.
* He's had an organ transplant.
* HIV infection, hepatitis C (hepatitis C antibody positive with HCV-RNA above the detection limit of the assay), chronic active hepatitis B (HBV DNA≥2×103IU/ml or >1×104copies/mL).
* Active tuberculosis, interstitial pneumonia, active infection, poorly controlled diabetes, symptomatic arrhythmia, symptomatic new dysfunction, myocardial infarction, active peptic ulcer, chronic active enteritis within 6 months; Affected during pregnancy or lactation.
* Major surgery in the last three months.
* Severe diabetes mellitus with poor drug control, symptomatic arrhythmia, symptomatic cardiac insufficiency, myocardial infarction within 6 months, chronic active enteritis, chronic nephritis. QTc acuity 470 ms.
* He had a history of malignancy. Previously received chemotherapy, radiotherapy, targeted therapy, immunotherapy and other antitumor therapies.
* Patients with allergic or contraindicated taxa.
* Live vaccine is administered within 30 days before the first dose of immunotherapy.
* Refusal or inability to sign up for ICF study.
* The investigator decided that the patient was not suitable to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete pathological response rate | 1 year

SECONDARY OUTCOMES:
R0 resection rate | 1 year
2-year Disease-free survival rate | 2 years
2-year overall survival rate | 2 years
Safety will be analyzed through the incidence of adverse events, serious adverse events | Up to 28 days from last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No